CLINICAL TRIAL: NCT04407312
Title: Adjunctive Cilostazol to Dual Antiplatelet Therapy to Enhance Mobilization of Endothelial Progenitor Cell in Patients With Acute Myocardial Infarction: A Randomized, Placebo-controlled ACCEL-EPISODE Trial
Brief Title: Cilostazol and Endothelial Progenitor Cell
Acronym: EPISODE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gyeongsang National University Hospital (Other)
Collaborators: Korea Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yongwhi Park, MD, PhD., Principal investigator, Gyeongsang National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GNUHIRB 2012-01-005
Record Dates: First submitted 2020-05-20; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Myocardial Infarction, Acute
Keywords: Endothelial progenitor cell; Myocardial infarction, acute; Platelets; Cilostazol
MeSH Terms: conditions — Myocardial Infarction | interventions — Cilostazol; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CILO group (Experimental): Intervention:
  Suspected patients with AMI were loaded with 600-mg clopidogrel and 300-mg aspirin in the emergency room.
  After 3 to 5 days post-PCI (before discharge), patients were randomly allocated to the CILO group or the placebo group (1:1 fashion) based on a computer-generated randomization sequence.
  For the CILO group, cilostazol-SR 200 mg daily was added to dual antiplatelet therapy with aspirin (100 mg daily) and clopidogrel (75 mg daily).
  Study drug is maintained for 30 days. Double blinded, Randomized, Placebo controlled Trial.
  Drug:
  Cilostazol-SR, Tablet, 200mg, once daily. Astrix, Capsule, 100mg, once daily. Plavix, tablet, 75mg, once daily.
  Interventions: Drug: Cilostazol Tablets; Drug: Aspirin; Drug: Clopidogrel
- Placebo group (Placebo Comparator): Intervention:
  Suspected patients with AMI were loaded with 600-mg clopidogrel and 300-mg aspirin in the emergency room.
  After 3 to 5 days post-PCI (before discharge), patients were randomly allocated to the CILO group or the placebo group (1:1 fashion) based on a computer-generated randomization sequence.
  In the Placebo group, placebo tablet was administered on top of dual antiplatelet therapy with aspirin (100 mg daily) and clopidogrel (75 mg daily).
  Study drug is maintained for 30 days. Double blinded, Randomized, Placebo controlled Trial.
  Drug:
  Placebo, Tablet, 200mg, once daily. Astrix, Capsule, 100mg, once daily. Plavix, tablet, 75mg, once daily.
  Interventions: Drug: placebo; Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Drug: Cilostazol Tablets — Cilostazol-SR, capsule, 200mg, once daily, 30 days.
  Other Names: Cilostazol-SR
  Arms: CILO group
Drug: placebo — Placebo, tablet, 200mg, once daily, 30 days.
  Arms: Placebo group
Drug: Aspirin — Astrix, capsule,100mg, once daily, 30 days.
  Other Names: Astrix
Drug: Clopidogrel — Plavix, tablet, 75mg, once daily, 30 days.
  Other Names: Plavix

SUMMARY:
To assess impact of adjunctive cilostazol on endothelial progenitor cell (EPC) mobilization in patients with acute myocardial infarction (To reveal the role of cilostazol in up-regulation of EPC count)

DETAILED DESCRIPTION:
Primary endpoint: % Change of EPC count

Secondary endpoints:

1. Changes of ADP/AA/collagen-induced PFT
2. Changes of lipid profile and high sensitivity-C-reactive protein
3. Change of TEG measurements
4. Change of PWV
5. Predictors of EPC count (baseline and 1-month)
6. ischemic (CV death, MI & stroke) and bleeding events (BARC)

ELIGIBILITY:
Inclusion Criteria:

* naïve AMI
* undergoing successful coronary stent implantation

Exclusion Criteria:

* high-risk patients for thrombotic event;
* a history of active bleeding or bleeding diatheses;
* contraindication to antiplatelet therapy;
* hemodynamic or electrical instability;
* oral anticoagulation therapy;
* left ventricular ejection fraction < 30%;
* leukocyte count < 3,000/mm3 and/or platelet count < 100,000/mm3;
* AST or ALT > 3 times the respective the upper limit;
* serum creatinine level > 3.5 mg/dL;
* stroke within 3 months;
* pregnancy;
* non-cardiac disease with a life expectancy < 1 year;
* any patients not tolerable or suitable for coronary intervention; and
* inability to follow the protocol

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline CD133+/KDR+ at 30 days | baseline and 30 days
  Peripheral blood mononuclear cells measurement by flow cytometry
Changes from baseline CD34+/KDR+ at 30 days | baseline and 30 days
  Peripheral blood mononuclear cells measurement by flow cytometry

SECONDARY OUTCOMES:
Levels of Platelet inhibition | baseline and 30 days
  Platelet function test by VerifyNow assay at 30-day follow-up
Correlation between the changes of CD133+/KDR+ and platelet reactivity unit by VerifyNow by Pearson's method | baseline and 30 days
  the correlation between the changes of EPC subsets and ∆Platelet reactivity unit (PRU) by Pearson's method
Correlation between the changes of CD34+/KDR+ and platelet reactivity unit by VerifyNow | baseline and 30 days
  the correlation between the changes of EPC subsets and ∆PRU by Pearson's method
Incidence of bleeding events by BACR definition | 30 days
  Safety outcome

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoon Jeong, MD,.PhD, Principal Investigator — Gyeongsang National University Changwon Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park Y, Kim JH, Kim TH, Koh JS, Hwang SJ, Hwang JY, Jeong YH. Adjunctive Cilostazol to Dual Antiplatelet Therapy to Enhance Mobilization of Endothelial Progenitor Cell in Patients with Acute Myocardial Infarction: A Randomized, Placebo-Controlled EPISODE Trial. J Clin Med. 2020 Jun 1;9(6):1678. doi: 10.3390/jcm9061678. PMID 32492942